CLINICAL TRIAL: NCT04589143
Title: Agomelatine Augmentation in Early-Nonresponsive Patients With Major Depressive Disorder Receiving SSRIs or SNRIs: a Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: A Double-blind, Placebo-controlled Study of Antidepressant Augmentation With Agomelatine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Lingjiang Li, President of Chinese Psychiatry Society of Chinese Medical Association, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Second Xiangya hospital
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: agomelatine; antidepressant; augmentation; major depressive disorder; early-nonresponsive
MeSH Terms: conditions — Depressive Disorder, Major | interventions — agomelatine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experience group (Experimental): In this group,participants take agomelatine at a dose of 25-50 mg/d for 8 weeks.
  Interventions: Drug: Agomelatine
- Contral group (Placebo Comparator): In this group,participants take a placebo at a dose of 25-50 mg/d for 8 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Agomelatine — Oral tablets of agomelatine at a dose of 25-50 mg/d for 8 weeks
  Arms: Experience group
Drug: Placebos — Oral tablets of placebos at a dose of 25-50 mg/d for 8 weeks
  Arms: Contral group

SUMMARY:
The purpose of this study was to investigate the efficacy and safety of antidepressant augmentation with agomelatine in the treatment of patients with depression who did not demonstrate satisfying response to selective serotonin reuptake inhibitor (SSRI) and serotonin-noradrenaline reuptake inhibitor (SNRI) during their early phase of treatment; this study also aims to explore the effects of augmenting antidepressant treatment with agomelatine on various aspects, including sleep quality, quality of life, social functioning, and cognitive function in patients with MDD.

ELIGIBILITY:
1. Age between 18 and 60 years.
2. Meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for a current major depressive episode.
3. Demonstrating an inadequate response to antidepressant treatment lasting at least 2 weeks, at the minimum effective dose for antidepressants. Inadequate response is defined as a < 20% change in the Hamilton Depression Rating Scale-17 (HAMD-17) score or as per patients' self-report in the antidepressant treatment questionnaire. Minimum effective doses for some commonly used classes of antidepressants include:

   * Sertraline: >50mg
   * Fluoxetine: >20 mg
   * Citalopram: >20 mg
   * Escitalopram: >10mg
   * Venlafaxine: >75 mg
   * Duloxetine: >50 mg
4. HAMD-17≥17; Clinical Global Impression-Severity (CGI-S) score ≥4.
5. Education level of at least 6 years, with the ability to independently complete all scales and assessments.
6. Agreement from primary healthcare providers and patients to maintain current antidepressant treatment while adding agomelatine.

**Exclusion Criteria:**

1. Meeting criteria for other psychiatric disorders according to DSM-IV (except generalized anxiety disorder), such as schizophrenia, bipolar disorder, or mental disorders related to alcohol and drug dependence.
2. Current or previous history of brain organic diseases or loss of consciousness for more than 5 minutes.
3. Current or previous history of major physical diseases (including rheumatic immune system diseases, endocrine and metabolic diseases, nervous system diseases, etc.).
4. Current serious suicidal ideation or suicide attempt.
5. Pregnancy or lactation in women.
6. Color blindness (which would hinder neurocognitive testing).
7. Use of anticoagulants (e.g., heparin, warfarin), glucocorticoids, or treatment for thyroid diseases in the past 3 months.
8. Having received any neurocognitive assessment similar to this study in the past 12 months.
9. Positive urine drug screening results or abnormal thyroid function test.
10. Liver function tests showing transaminase (ALT and AST) levels 2 times above the upper limit of the normal range.
11. Electrocardiogram examination revealing a QTc ≥ 430 ms in males or QTc ≥ 450 ms in females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 137 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale scores | Baseline (week 0), week 2, week 4, week 8
  Depression severity; higher scores mean a worse outcome.
Side Effect Rating Scale (SERS) scores | Baseline (week 0), week 2, week 4, week 8
  Safety: frequency and severity of adverse events; higher scores mean a better outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) scores | Baseline (week 0), week 2, week 4, week 8
  Self-report depression severity; higher scores mean a worse outcome.
Hamilton Anxiety Rating Scale (HAMA) scores | Baseline (week 0), week 2, week 4, week 8
  Anxiety severity; higher scores mean a worse outcome.
General Anxiety Disorder-7 (GAD-7) scores | Baseline (week 0), week 2, week 4, week 8
  Self-report anxiety severity; higher scores mean a worse outcome.
Changes in Clinical Global Impression (CGI) scores | Baseline (week 0), week 2, week 4, week 8
  Symptom severity; higher scores mean a worse outcome.
Snaith-Hamilton Pleasure Scale (SHAPS) scores | Baseline (week 0), week 2, week 4, week 8
  Self-reported severity of anhedonia; higher scores mean a worse outcome.
Sheehan Disability Scale (SDS) scores | Baseline (week 0), week 2, week 4, week 8
  Self-report tool that assesses functional impairment in work/school, social life, and family life; higher scores mean a worse outcome.
Quality of life (EQ-5D-3L) scores | Baseline (week 0), week 2, week 4, week 8
  Self-report Quality of life; higher scores mean a better outcome.
performance of Neurocognitive test, including executive function, attention, processing speed, and memory | Baseline (week 0), week 2, week 4, week 8
  Neurocognitive function; higher scores mean a better outcome.
Athens Insomnia Scale (AIS) scores | Baseline (week 0), week 2, week 4, week 8
  Self-report severity of insomnia; higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute & Faculty of Psychiatry of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ju Y, Ou W, Chen H, Yang L, Long Y, Liang H, Xi Z, Huang M, Chen W, Lv G, Shao F, Liu B, Liu J, Li Z, Liao M, Liang W, Yao Z, Zhang Y, Li L. Agomelatine as adjunctive therapy with SSRIs or SNRIs for major depressive disorder: a multicentre, double-blind, randomized, placebo-controlled trial. BMC Med. 2025 Mar 5;23(1):137. doi: 10.1186/s12916-025-03951-0. PMID 40038707